CLINICAL TRIAL: NCT03425240
Title: Intra-operative Neuromodulation of the Pelvic Plexus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laikο General Hospital, Athens (Other)
Responsible Party: Principal Investigator, Dr. Ioannis Adamakis, MD, Principal investigator, Laikο General Hospital, Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 7818
Record Dates: First submitted 2018-01-24; First posted 2018-02-07 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Erectile Dysfunction; Prostate Cancer
Keywords: Erectile Dysfunction; Prostate Cancer; Neuromodulation
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nerve Stimulation (Experimental): Acute placement of electrodes and electrostimulation of the pelvic plexus nerves during open radical prostatectomy.
  Interventions: Device: Nerve Stimulation

INTERVENTIONS:
Device: Nerve Stimulation — Acute placement of electrodes on the pelvic plexus to apply electrostimulation during open radical prostatectomy.

SUMMARY:
The purpose of this study is to evaluate the feasibility of electrical stimulation of nerves responsible for erectile function to evoke penile erection after surgery to remove the prostate (prostatectomy).

DETAILED DESCRIPTION:
Prostate cancer is the main cancer in men. However, the survival rate for clinically localized prostate cancer is prominent mainly due to radical prostatectomy (RP), the gold standard treatment for non-metastatic cancers. Unfortunately, despite providing optimal cancer control, RP often lead to neuropraxia and persistent erectile dysfunction in approximately 80% of men 1 year after prostatectomy. Various erectile rehabilitation strategies have not been able to prove a beneficial action yet. However, electrical stimulation has been demonstrated to favour neuroregeneration and the functional recovery of neuromuscular systems and has been shown to induce and maintain penile erection in animals and humans. Therefore, electrical stimulation of the pelvic plexus nerves during radical prostatectomy is being investigated for its potential development into a treatment aimed at improving recovery of erectile function after prostatectomy.

The primary objective of this study is to explore the feasibility of using a neurostimulation device post radical prostatectomy as a method for neurogenic erectile dysfunction treatment. During standard open radical prostatectomy, the pelvic plexus nerves will be electrically stimulated intraoperatively and the modification of penile circumference will be recorded.

The secondary objective is to assess proper placement of the stimulation electrodes and stimulation parameters needed to achieve maximal change in penile circumference.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for open radical prostatectomy procedure under total anesthesia.
* Age 40 to 75 years old.
* Able to read and understand patient information materials and willing to sign a written informed consent.

Exclusion Criteria:

* Have been diagnosed with severe vasculogenic erectile dysfunction.
* Have a prior history of pelvic surgery, trauma or irradiation therapy.
* Have a penile prosthesis.
* Have been diagnosed with neurologic diseases that may negatively impact erectile functions.
* Currently having an active implantable device (such as a pacemaker).
* Posses any other characteristics that, per the investigator's judgment, may increase the risk or impair data collection for the procedure/study.
* Inability to provide a fully informed consent.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-09-10 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Penile circumference increase in millimeters. | 5 minutes
  Change in penile circumference [mm] in response to electrical stimulation of the pelvic plexus nerves measured by a penile plethysmograph.

SECONDARY OUTCOMES:
Anatomic location of stimulation site | 5 to 15 minutes
  The anatomic location of the stimulation site on the pelvic floor (determined by the surgeon).
Stimulation threshold in volts | 5 to 15 minutes
  Amplitude in volts of the electrical stimulation pulses to induce penile response.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Adamakis, MD, Principal Investigator — Laikon General Hospital of Athens; Constantinos A. Constantinides, MD, Study Chair — Laikon General Hospital of Athens
Locations (1):
- Laikon General Hospital of Athens, Athens, Greece